CLINICAL TRIAL: NCT05542966
Title: Blender Biomarkers: A BLENDER Sub-study to Evaluate the Effect of Oxygen Dose on Oxidative Stress and Organ Injury
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: HREC/50486/Alfred-2019
Record Dates: First submitted 2022-04-13; First posted 2022-09-16 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Failure; Critical Illness
Keywords: ECMO; V-A ECMO; Oxidative stress; Oxygen; Hyperoxia
MeSH Terms: conditions — Heart Failure; Critical Illness; Hyperoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To compare the impact of liberal vs conservative oxygen doses on markers of oxidative stress in patients enrolled in the BLENDER trial.

DETAILED DESCRIPTION:
Extracorporeal membrane oxygen (ECMO) is a heart lung support device used for patients with severe and cardiac and respiratory failure and carries an increased risk of exposure to very high oxygen tensions. Hyperoxia (arterial oxygen >100mmHg) can lead to the production of reactive oxygen species (ROS). Excess production of ROS and depletion of antioxidant compounds is referred to as oxidative stress and results in inflammation, tissue injury and cell death. The inter-relationship between the production of ROS and end organ dysfunction is complicated and remain unclear. A more detailed assessment of the timing of changes in markers of oxidative stress, inflammatory mediators and tissue injury is warranted to understand the processes and potentially identify therapeutic targets.

The BLENDER Trial is a multicentre trial in ECMO patients to determine whether a conservative oxygen strategy during ECMO reduces ICU length of stay and improves patient outcomes compared to a liberal oxygen strategy. Currently there have been no studies that look at the underlying pathophysiological changes that occur in patients on ECMO when subjected to different oxygen concentrations. As such The BLENDER study represents a unique opportunity to understand the mechanisms by which hyperoxia may cause tissue injury in patients receiving ECMO. This nested study seeks to elucidate whether exposure to hyperoxia during ECMO results in increased oxidative stress and whether this is correlated with increased risk of tissue injury and organ dysfunction. A better understanding of the mechanism of hyperoxia induced tissue injury may allow treatment to be optimised for patients exposed to hyperoxia as part of their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving venoarterial (VA) ECMO
* Enrolled in the BLENDER trial

Exclusion Criteria:

* Not enrolled in the BLENDER trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: VA-ECMO patients enrolled in the BLENDER trial
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Super oxide dismutase levels U/ml | Within 24 hours of ECMO commencement
  Plasma levels of superoxide dismutase in patients exposed to either a liberal or conservative oxygen strategy during VA-ECMO

SECONDARY OUTCOMES:
Marker of Cardiac Injury | Day 3 of ECMO
  Troponin ng/ml
  This will be determined by analysing blood samples routinely collected daily from patient receiving ECMO
Marker of Cardiac Injury | Day 7 of ECMO
  Troponin I ng/ml
  This will be determined by analysing blood samples routinely collected daily from patient receiving ECMO
Markers of Liver Injury | Day 3 of ECMO
  ALT and AST (IU/L)
  This will be determined by analysing blood samples routinely collected daily from patient receiving ECMO
Markers of Liver Injury | Day 7 of ECMO
  ALT and AST (IU/L)
  This will be determined by analysing blood samples routinely collected daily from patient receiving ECMO
Marker of Neurological Injury | Day 3 of ECMO
  Neuron Specific Enolase (microg/L)
  This will be determined by analysing blood samples routinely collected daily from patient receiving ECMO
Marker of Neurological Injury | Day 7 of ECMO
  Neuron Specific Enolase (microg/L)
  This will be determined by analysing blood samples routinely collected daily from patient receiving ECMO
Coagulation Parameters | Day 3 of ECMO
  APTT
  This will be determined by analysing blood samples routinely collected daily from patient receiving ECMO
Coagulation Parameters | Day 7 of ECMO
  APTT
  This will be determined by analysing blood samples routinely collected daily from patient receiving ECMO
Immune Markers | Day 3 of ECMO
  IL-6, TNFa, IL-10, IL-1B (pg/ml)
Immune Markers | Day 7 of ECMO
  IL-6, TNFa, IL-10, IL-1B (pg/ml)
Other Markers of Oxidative Stress | Day 3 of ECMO
  Malondialdehyde, Vitamin C
Other Markers of Oxidative Stress | Day 7 of ECMO
  Malondialdehyde, Vitamin C
Superoxide dismutase levels U/ml | On Day 3 following ECMO commencement
  Plasma levels of superoxide dismutase in patients exposed to either a liberal or conservative oxygen strategy during VA-ECMO
Superoxide dismutase levels | On Day 7 following ECMO commencement
  Plasma levels of superoxide dismutase in patients exposed to either a liberal or conservative oxygen strategy during VA-ECMO
Markers of Kidney Injury | Day 3 of ECMO
  Creatinine (micromol/L)
Markers of Kidney Injury | Day 7 of ECMO
  Creatinine (micromol/L)

OTHER OUTCOMES:
Marker of Fibrinolysis | Day 3 of ECMO
  Fibrinogen, Plasmin anti-plasmin complex, D-Dimer
  This will be determined by analysing blood samples routinely collected daily from patient receiving ECMO
Marker of Fibrinolysis | Day 7 of ECMO
  Fibrinogen, Plasmin anti-plasmin complex, D-dimer
  This will be determined by analysing blood samples routinely collected daily from patient receiving ECMO

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided